CLINICAL TRIAL: NCT06359639
Title: Randomised Controlled Trial of Cognitive Restructuring in Managing Breakup Distress and Promoting Posttraumatic Growth
Brief Title: Cognitive Restructuring in Managing Breakup Distress and Promoting Posttraumatic Growth Among Malaysian Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Choong Poh Kin (Other)
Responsible Party: Sponsor-Investigator, Michelle Choong Poh Kin, Doctor of Clinical Psychology candidate, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/23080645
Record Dates: First submitted 2024-03-09; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Breakup Distress; Posttraumatic Growth
MeSH Terms: interventions — Cognitive Restructuring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive restructuring (Experimental)
  Interventions: Behavioral: Cognitive restructuring
- Supportive counselling (Active Comparator)
  Interventions: Behavioral: Supportive counselling

INTERVENTIONS:
Behavioral: Cognitive restructuring — Five 50-60-minute videoconferencing sessions of cognitive restructuring based on Mind Over Mood: Second Edition (MOM2) (Greenberger & Padesky, 2016) and The Clinician's Guide to CBT Using MOM2 (Padesky & Greenberger, 2019) as guides. The sessions will consist of understanding the cognitive model, filling in Thought Records, and complementary coping strategies of looking for evidence, action planning, and acceptance.
  Arms: Cognitive restructuring
Behavioral: Supportive counselling — Five 50-60-minute videoconferencing sessions of supportive counselling consisting of psychoeducation on breakup effects, validation of breakup experiences and emotions, introduction to deep breathing and progressive muscle relaxation, and identification of existing coping strategies.
  Arms: Supportive counselling

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of cognitive restructuring in reducing breakup distress and promoting personal growth among Malaysian young adults. Cognitive restructuring is a therapy skill that focuses on changing unhelpful thoughts. The main question it aims to answer is: Are there differences in their breakup distress and personal growth after receiving cognitive restructuring compared to counselling? Participants will receive five online sessions of either cognitive restructuring or counselling. Data on participants' breakup distress and personal growth will be collected before and after completion of sessions. The hypothesis is that cognitive restructuring will reduce breakup distress and increase personal growth more than counselling.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian young adults.
* Proficient in English.
* Basic technological skill and resources.
* Reported ongoing distress due to a breakup that occurred within the past 6 months.
* Current single relationship status.

Exclusion Criteria:

* Consumption of psychiatric medications within past 8 weeks.
* Currently receiving other psychological interventions.
* Presence of significant psychotic or manic symptoms.
* Severe suicide risk.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Breakup distress | BDS will be administered: 1) before the start of intervention sessions, 2) after 5 weeks of intervention sessions, and 3) 1 month after the participant's 5th (final) intervention session.
  Breakup Distress Scale (BDS) (Field et al., 2009) will be used to assess breakup distress. The total score ranges from 16 to 64 with higher scores indicating higher breakup distress.
Posttraumatic growth | PTGI will be administered: 1) before the start of intervention sessions, 2) after 5 weeks of intervention sessions, and 3) 1 month after the participant's 5th (final) intervention session.
  Posttraumatic Growth Inventory (PTGI) (Tedeschi & Calhoun, 1996) will be used to assess personal growth after breakup. The total score ranges from 0 to 105 with higher scores indicating higher posttraumatic growth.

IPD SHARING:
Plan to Share IPD: No